CLINICAL TRIAL: NCT04211727
Title: Affinity: Hospital Trial. Early Prototype Testing for a Home Oncology Monitoring System
Brief Title: Affinity: Hospital Trial
Status: Completed | Type: Observational
Sponsor: Entia Ltd (Industry)
Collaborators: The Christie NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: IRAS ID 275879
Record Dates: First submitted 2019-12-18; First posted 2019-12-26 (Actual); Last update posted 2022-03-29 (Actual); Status verified 2022-03

CONDITIONS: Cancer
Keywords: Oncology; Cancer
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cohort 1: Patients receiving standard of care systemic anti-cancer therapy for solid organ malignancy and has received at least one cycle aged 18 years and over.
  Interventions: Diagnostic Test: Capillary finger prick blood sample
- Cohort 2: Patients receiving standard of care systemic anti-cancer therapy for solid organ malignancy and has received at least one cycle aged 18 years and over.
  Interventions: Diagnostic Test: Capillary finger prick blood sample

INTERVENTIONS:
Diagnostic Test: Capillary finger prick blood sample — Patients will have a blood finger prick sample

SUMMARY:
Method comparison study to compare the Affinity prototype device using a capillary blood sample against routine venous laboratory results, in patients undergoing systemic anti-cancer therapy (SACT). Tests will be performed by healthcare professionals (Cohort 1) and participants self-testing (Cohort 2)

DETAILED DESCRIPTION:
In this study the Investigators wish to compare 200 finger prick sample (capillary) blood results taken and analysed using the Affinity prototype device to standard of care venous blood samples, taken from the participant on the same day. The blood tests will analyse Full Blood Count (FBC)

200 patients will be recruited in total. 100 will take part in Cohort 1, where a member of the clinical research team will take their blood sample using the Affinity prototype device. The other 100 will take part in Cohort 2, where the participant will self test and take the blood sample themselves. Participants will be asked to complete a short questionnaire after using the device to provide any feedback on its design and use.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years old at the time of study entry Currently receiving standard of care systemic anti-cancer therapy for solid organ malignancy and has received at least one cycle
* Scheduled to be undergoing routine venous laboratory blood tests as part of standard of care
* Can provide written informed consent
* Cohort 2 only- Able to independently complete participant questionnaires

Exclusion Criteria:

* Receiving systemic anti-cancer therapy for a haematological malignancy
* Known parasitic infection
* Known inherited or acquired bleeding disorder
* History of haematological malignancy
* Known poorly controlled anti-coagulation
* Cohort 2 only- Participant or carer unable or unlikely to be able to perform fine manipulation required to use lancet or cartridge to obtain capillary blood sample and result

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing systemic anti-cancer therapy (SACT)
Sampling Method: Non-Probability Sample
Enrollment: 247 (Actual)
Dates: Start 2020-10-26 (Actual); Primary Completion 2022-01-17 (Actual); Study Completion 2022-01-17 (Actual)

PRIMARY OUTCOMES:
To assess the accuracy (bias) of the Affinity prototype device against laboratory testing (capillary vs. venous sample) | 1 year
  Measuring Full Blood Count (FBC)

SECONDARY OUTCOMES:
Assessment and feedback | 1 year
  To measure the number of issues when the prototype device is used by healthcare professionals (Cohort 1) and participants (Cohort 2).
Assessment and feedback | 1 year
  To measure the severity of each issue when the prototype device is used by healthcare professionals (Cohort 1) and participants (Cohort 2).

CONTACTS AND LOCATIONS:
Locations (1):
- The Christie NHS Foundation Trust, Manchester, United Kingdom

IPD SHARING:
Plan to Share IPD: No